CLINICAL TRIAL: NCT06507605
Title: Phase 1 Randomized, Double-blind Dose-Escalating Study of Pfs230D1 in Combination With R21 in Matrix-M in Healthy African Adults
Brief Title: Dose-Escalating Study of Pfs230D1 in Combination With R21 in Matrix-M in African Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VIMT 001
Record Dates: First submitted 2024-07-04; First posted 2024-07-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Prevention of Malaria Transmission and Clinical Malaria
MeSH Terms: interventions — R21 monoclonal antibody; Matrix-M

STUDY DESIGN:
Intervention Model Description: Participants will be randomized by cohorts as to one of the study arms to receive single antigen (Pfs230D1 or R21) or combination (Pfs230D1 + R21) with 50 μg of Matrix-M, all administered as an IM injection on a 1, 29, 57-day schedule.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Arm 1a (n=20) (Experimental): 6μg Pfs230D1-CRM197 + 5μg of R21 in 50μg Matrix-M
  Interventions: Biological: R21; Biological: Pfs230D1-CRM197; Other: Matrix-M
- Arm 1b (n=20) (Experimental): 6μg Pfs230D1-CRM197 + 10μg of R21 in 50μg Matrix-M
  Interventions: Biological: R21; Biological: Pfs230D1-CRM197; Other: Matrix-M
- Arm 1c (n=20) (Experimental): 12μg Pfs230D1-CRM197 + 5μg of R21 in 50μg Matrix-M
  Interventions: Biological: R21; Biological: Pfs230D1-CRM197; Other: Matrix-M
- Arm 1d (n=20) (Experimental): 12μg Pfs230D1-CRM197 + 10μg of R21 in 50μg Matrix-M
  Interventions: Biological: R21; Biological: Pfs230D1-CRM197; Other: Matrix-M
- Arm 1e (n=20) (Active Comparator): 5μg of R21 in 50μg Matrix-M
  Interventions: Biological: R21; Other: Matrix-M
- Arm 1f (n=20) (Active Comparator): 10μg of R21 in 50μg Matrix-M
  Interventions: Biological: R21; Other: Matrix-M
- Arm 2a (n=20) (Experimental): 20μg Pfs230D1-CRM197 + 5μg of R21 in 50μg Matrix-M
  Interventions: Biological: R21; Biological: Pfs230D1-CRM197; Other: Matrix-M
- Arm 2b (n=20) (Experimental): 20μg Pfs230D1-CRM197 + 10μg of R21 in 50μg Matrix-M
  Interventions: Biological: R21; Biological: Pfs230D1-CRM197; Other: Matrix-M
- Arm 2c (n=20) (Experimental): 20μg Pfs230D1-CRM197 in 50μg Matrix-M
  Interventions: Biological: Pfs230D1-CRM197; Other: Matrix-M
- Arm 2d (n=20) (Experimental): 20μg Pfs230D1-EPA + 5μg of R21 in 50μg Matrix-M
  Interventions: Biological: R21; Biological: Pfs230D1-EPA; Other: Matrix-M
- Arm 3a (n=20) (Experimental): 40μg Pfs230D1-CRM197 + 5μg of R21 in 50μg Matrix-M
  Interventions: Biological: R21; Biological: Pfs230D1-CRM197; Other: Matrix-M
- Arm 3b (n=20) (Experimental): 40μg Pfs230D1-CRM197 + 10μg of R21 in 50μg Matrix-M
  Interventions: Biological: R21; Biological: Pfs230D1-CRM197; Other: Matrix-M

INTERVENTIONS:
Biological: R21 — R21 is a portion of Pf circumsporozoite protein fused with hepatitis B surface antigen in the form of non-infectious virus-like particles (VLPs) produced in yeast cells (Hansenula) by recombinant DNA technology.
  Arms: Arm 1a (n=20); Arm 1b (n=20); Arm 1c (n=20); Arm 1d (n=20); Arm 1e (n=20); Arm 1f (n=20); Arm 2a (n=20); Arm 2b (n=20); Arm 2d (n=20); Arm 3a (n=20); Arm 3b (n=20)
Biological: Pfs230D1-CRM197 — Recombinant Pfs230 domain 1 (Pfs230D1; a subdomain of a surface antigen of gametocytes, gametes, and zygotes, in the mosquito stage of Pf conjugated to CRM197 and adjuvanted with 50μg of Matrix-M.
  Arms: Arm 1a (n=20); Arm 1b (n=20); Arm 1c (n=20); Arm 1d (n=20); Arm 2a (n=20); Arm 2b (n=20); Arm 2c (n=20); Arm 3a (n=20); Arm 3b (n=20)
Biological: Pfs230D1-EPA — Recombinant Pfs230D1 conjugated to a recombinant Pseudomonas aeruginosa ExoProtein A (EPA)
  Arms: Arm 2d (n=20)
Other: Matrix-M — Vaccine adjuvant that contains purified saponin (from Quillaja saponaria Molina) and cholesterol and phosphatidyl choline. Matrix-M will be used at a 50μg dose for vaccinations.

SUMMARY:
This is a Phase 1, individually randomized, double-blind, dose escalating study designed to evaluate the safety, tolerability, and immunogenicity of Pfs230D1 conjugate vaccines, R21 nanoparticle vaccine, or their combination conjugate vaccines, formulated on Matrix-M in healthy African adults aged 18 to 50 years.

DETAILED DESCRIPTION:
240 healthy adults (18-50 years of age) will be enrolled from Mali, Africa in a staggered manner by increasing Pfs230D1 dosing.

Participants will be randomized by cohorts as (detailed below) to one of the study arms to receive single antigen (Pfs230D1 or R21) or combination (Pfs230D1 + R21) with 50 μg of Matrix-M, all administered as an IM injection on a 1, 29, 57-day schedule. Participants will be followed for safety for 6 months post last dose with continued assessment for clinical malaria cases and immunogenicity up until 12 months post last dose.

Cohort 1 (n=120); 1:1:1:1:1:1

* Arm 1a (n=20): 6μg Pfs230D1-CRM197 + 5μg of R21 in 50μg Matrix-M
* Arm 1b (n=20): 6μg Pfs230D1-CRM197 + 10μg of R21 in 50μg Matrix-M
* Arm 1c (n=20): 12μg Pfs230D1-CRM197 + 5μg of R21 in 50μg Matrix-M
* Arm 1d (n=20): 12μg Pfs230D1-CRM197 + 10μg of R21 in 50μg Matrix-M
* Arm 1e (n=20): 5μg of R21 in 50μg Matrix-M
* Arm 1f (n=20): 10μg of R21 in 50μg Matrix-M

Followed by Cohort 2 (n=80); 1:1:1:1

* Arm 2a (n=20): 20μg Pfs230D1-CRM197 + 5μg of R21 in 50μg Matrix-M
* Arm 2b (n=20): 20μg Pfs230D1-CRM197 + 10μg of R21 in 50μg Matrix-M
* Arm 2c (n=20): 20μg Pfs230D1-CRM197 in 50μg Matrix-M
* Arm 2d (n=20): 20μg Pfs230D1-EPA + 5μg of R21 in 50μg Matrix-M

Followed by Cohort 3 (n=40); 1:1

* Arm 3a (n=20): 40μg Pfs230D1-CRM197 + 5μg of R21 in 50μg Matrix-M
* Arm 3b (n=20): 40μg Pfs230D1-CRM197 + 10μg of R21 in 50μg Matrix-M

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 50 years old.
2. Provides written informed consent.
3. Able to understand and comply with planned study procedures and be available for the duration of the trial.
4. In good general health and without clinically significant medical history in the opinion of the investigator.
5. Females of childbearing potential must be willing to use reliable contraception from 21 days prior to Study Day 1 and until 1 month after the last vaccination.

Exclusion Criteria:

1. Pregnant and breastfeeding females.
2. Hemoglobin, white blood cell (WBC), absolute neutrophil count, or platelet levels outside the local laboratory-defined reference ranges.
3. Alanine transaminase (ALT) or creatinine (Cr) level above the local laboratory-defined upper limit of reference range.
4. Infected with HIV, hepatitis B, hepatitis C.
5. Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, hematological, oncologic, or renal disease by history, physical examination, and/or laboratory studies.
6. Current or planned participation in an investigational product study until the time period of the last required study visit under this protocol.
7. Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
8. History of a severe allergic reaction or anaphylaxis.
9. Known: Severe asthma, Autoimmune or antibody-mediated disease, Immunodeficiency, Seizure disorder, Asplenia or functional asplenia, Use of chronic oral or intravenous corticosteroids (excluding topical or nasal), Sickle cell disease.
10. Any other condition that in the opinion of the investigator might jeopardize the safety or rights of a subject participating in the trial, interfere with the evaluation of the study objectives, or might render the subject unable to comply with the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-01-24 (Actual); Study Completion 2026-01-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Immediate adverse events | within 30-minutes following each dose
  Occurrence of immediate adverse events
Number of Participants with Solicited local adverse events | for 7 days following each dose
  Occurrence of solicited local adverse events
Number of Participants with Solicited systemic adverse events | for 7 days following each dose
  Occurrence of solicited systemic adverse events
Number of Participants with Unsolicited adverse events | for 28 days following each dose
  Occurrence of all unsolicited adverse events
Number of Participants with Abnormal Laboratory Values post-vaccination | within 7 days following each dose
  Any significant change from baseline for laboratory values defined as adverse events
Number of Participants with Serious adverse events | Till 6 months post last dose
  Occurrence of serious adverse events

SECONDARY OUTCOMES:
Anti-NANP IgG antibodies | at 2 weeks post dose 3 in all treatment arms
  Comparison of anti-NANP IgG antibodies
Anti-Pfs230D1 IgG antibodies | at 2 weeks post dose 3 in all treatment arms
  Comparison of Anti-Pfs230D1 IgG antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- University of Science, Technique and Technology of Bamako (Usttb), Bamako, Mali

IPD SHARING:
Plan to Share IPD: No